CLINICAL TRIAL: NCT01477580
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Tetravalent Recombinant Subunit Dengue Vaccine (V180) in Healthy Adults
Brief Title: Study of a Dengue Vaccine (V180) in Healthy Adults (V180-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V180-001
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (13):
- Low-dose V180 with low-dose ISCOMATRIX™ adjuvant (Experimental)
  Interventions: Biological: Low-dose V180 with low-dose ISCOMATRIX™ adjuvant
- Low-dose V180 with medium-dose ISCOMATRIX™ adjuvant (Experimental)
  Interventions: Biological: Low-dose V180 with medium-dose ISCOMATRIX™ adjuvant
- Medium-dose Non-adjuvanted V180 (Experimental)
  Interventions: Biological: Medium-dose V180 (non-adjuvanted)
- Medium-dose V180 with low-dose ISCOMATRIX™ adjuvant (Experimental)
  Interventions: Biological: Medium-dose V180 with low-dose ISCOMATRIX™ adjuvant
- Medium-dose V180 with medium-dose ISCOMATRIX™ adjuvant (Experimental)
  Interventions: Biological: Medium-dose V180 with medium-dose ISCOMATRIX™ adjuvant
- Medium-Dose V180 with Alhydrogel™ adjuvant (Experimental)
  Interventions: Biological: Medium-dose V180 with Alhydrogel™ adjuvant
- High-dose Non-adjuvanted V180 (Experimental)
  Interventions: Biological: High-dose V180 (non-adjuvanted)
- High-dose V180 with low-dose ISCOMATRIX™ adjuvant (Experimental)
  Interventions: Biological: High-dose V180 with low-dose ISCOMATRIX™ adjuvant
- High-dose V180 with medium-dose ISCOMATRIX™ adjuvant (Experimental)
  Interventions: Biological: High-dose V180 with medium-dose ISCOMATRIX™ adjuvant
- Low-dose V180 with high-dose ISCOMATRIX™ adjuvant (Experimental)
  Interventions: Biological: Low-dose V180 with high-dose ISCOMATRIX™ adjuvant
- Medium-dose V180 with high-dose ISCOMATRIX™ adjuvant (Experimental)
  Interventions: Biological: Medium-dose V180 with high-dose ISCOMATRIX™ adjuvant
- High-dose V180 with high-dose ISCOMATRIX™ adjuvant (Experimental)
  Interventions: Biological: High-dose V180 with high-dose ISCOMATRIX™ adjuvant
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low-dose V180 with low-dose ISCOMATRIX™ adjuvant — Three 0.5-mL intramuscular doses of low-dose V180 containing low-dose ISCOMATRIX™ adjuvant at Months 0, 1, and 2
  Arms: Low-dose V180 with low-dose ISCOMATRIX™ adjuvant
Biological: Low-dose V180 with medium-dose ISCOMATRIX™ adjuvant — Three 0.5-mL intramuscular doses of low-dose V180 containing medium-dose ISCOMATRIX™ adjuvant at Months 0, 1, and 2
  Arms: Low-dose V180 with medium-dose ISCOMATRIX™ adjuvant
Biological: Medium-dose V180 (non-adjuvanted) — Three 0.5-mL intramuscular doses of medium-dose V180 with no adjuvant at Months 0, 1, and 2
  Arms: Medium-dose Non-adjuvanted V180
Biological: Medium-dose V180 with low-dose ISCOMATRIX™ adjuvant — Three 0.5-mL intramuscular doses of medium-dose V180 containing low-dose ISCOMATRIX™ adjuvant at Months 0, 1, and 2
  Arms: Medium-dose V180 with low-dose ISCOMATRIX™ adjuvant
Biological: Medium-dose V180 with medium-dose ISCOMATRIX™ adjuvant — Three 0.5-mL intramuscular doses of medium-dose V180 containing medium-dose ISCOMATRIX™ adjuvant at Months 0, 1, and 2
  Arms: Medium-dose V180 with medium-dose ISCOMATRIX™ adjuvant
Biological: Medium-dose V180 with Alhydrogel™ adjuvant — Three 0.5-mL intramuscular doses of medium-dose V180 containing Alhydrogel™ adjuvant at Months 0, 1, and 2
  Arms: Medium-Dose V180 with Alhydrogel™ adjuvant
Biological: High-dose V180 (non-adjuvanted) — Three 0.5-mL intramuscular doses of high-dose V180 with no adjuvant at Months 0, 1, and 2
  Arms: High-dose Non-adjuvanted V180
Biological: High-dose V180 with low-dose ISCOMATRIX™ adjuvant — Three 0.5-mL intramuscular doses of high-dose V180 containing low-dose ISCOMATRIX™ adjuvant at Months 0, 1, and 2
  Arms: High-dose V180 with low-dose ISCOMATRIX™ adjuvant
Biological: High-dose V180 with medium-dose ISCOMATRIX™ adjuvant — Three 0.5-mL intramuscular doses of high-dose V180 containing medium-dose ISCOMATRIX™ adjuvant at Months 0, 1, and 2
  Arms: High-dose V180 with medium-dose ISCOMATRIX™ adjuvant
Biological: Low-dose V180 with high-dose ISCOMATRIX™ adjuvant — Three 0.5-mL intramuscular doses of low-dose V180 containing high-dose ISCOMATRIX™ adjuvant at Months 0, 1, and 2
  Arms: Low-dose V180 with high-dose ISCOMATRIX™ adjuvant
Biological: Medium-dose V180 with high-dose ISCOMATRIX™ adjuvant — Three 0.5-mL intramuscular doses of medium-dose V180 containing high-dose ISCOMATRIX™ adjuvant at Months 0, 1, and 2
  Arms: Medium-dose V180 with high-dose ISCOMATRIX™ adjuvant
Biological: High-dose V180 with high-dose ISCOMATRIX™ adjuvant — Three 0.5-mL intramuscular doses of high-dose V180 containing high-dose ISCOMATRIX™ adjuvant at Months 0, 1, and 2
  Arms: High-dose V180 with high-dose ISCOMATRIX™ adjuvant
Biological: Placebo — Three 0.5-mL intramuscular doses of phosphate-buffered saline at Months 0, 1, and 2
  Arms: Placebo

SUMMARY:
This study will determine whether at least one formulation of an experimental dengue vaccine (V180) is safe and causes an immune response.

ELIGIBILITY:
Selected Inclusion Criteria:

* In good health
* Voluntarily agrees to participate by giving written informed consent
* Able to read, understand, and complete study questionnaires
* Able to complete all scheduled visits and comply with study procedures
* Access to a telephone
* Agrees to avoid unusual, vigorous exercise from 72 hours before any dose of study vaccine/placebo through 15 days after that dose
* Weighs ≥110 pounds (50 kg) and has a body mass index (BMI) of 19 to 32 kg/m^2
* No fever (temperature ≥100.4°F/38.0°C) for 72 hours prior to vaccination
* Females of reproductive potential agree to remain abstinent or to use 2 acceptable methods of birth control from enrollment through 6 weeks after the last dose of study vaccine/placebo

Selected Exclusion Criteria:

* History of receiving any flavivirus vaccine (e.g. Japanese encephalitis, tick-borne encephalitis, or yellow fever) or planned receipt of any such vaccine during the study period
* History of any flavivirus infection or serologic evidence of any flavivirus infection, including West Nile, dengue, yellow fever, Saint Louis encephalitis (if available), Kunjin, Murray Valley encephalitis, and Japanese encephalitis
* History of residence for a cumulative period of >1 year in a country where dengue, Japanese encephalitis virus, or yellow fever virus is common
* Planned travel to an area where dengue is common through 28 days after receiving the last dose of study vaccine/placebo
* Known hypersensitivity to any component of the dengue vaccine
* Abuse of drugs or alcohol within 12 months prior to screening
* Pregnant or breastfeeding, or expecting to conceive in the time from enrollment through 6 weeks after the last dose of study vaccine/placebo
* Positive serum test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), and/or hepatitis C antibody
* Known, suspected, or a history of immunocompromise
* History of malignancy within 5 years prior to enrollment
* Poorly controlled diabetes mellitus
* Use of any immunosuppressive therapy (except topical and inhaled/nebulized steroids)
* Receipt of any licensed non-live vaccine within 14 days prior to the first dose of study vaccine/placebo or plans to receive a licensed non-live vaccine during the time between receiving the first dose and 28 days after receiving the last dose of study vaccine/placebo
* Receipt of any licensed live vaccine within 30 days prior to the first dose of study vaccine/placebo or plans to receive a licensed live vaccine during the time between receiving the first dose and 28 after receiving the last dose of study vaccine/placebo
* Received investigational drugs or vaccines within 2 months prior to the first dose of study vaccine/placebo
* History of receiving 1 or more doses of an investigational dengue vaccine
* Participation in another clinical study within 42 days prior to enrollment, or plans to participate in another clinical study from enrollment through 1 year after the last dose of study vaccine/placebo
* Planned donation of eggs or sperm from the time of enrollment through 28 days after the last dose of study vaccine/placebo
* Prior receipt of a blood transfusion or blood products within 6 months prior to the first dose of study vaccine/placebo
* Hospitalization for acute illness within 3 months prior to the first dose of vaccine/placebo

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2012-07-23 (Actual); Primary Completion 2014-01-23 (Actual); Study Completion 2014-12-11 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate for each serotype | 28 days postdose 3 (Day 84)
Geometric mean titer (GMT) of virus neutralizing antibodies for each serotype | 28 days postdose 3 (Day 84)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Manoff SB, Sausser M, Falk Russell A, Martin J, Radley D, Hyatt D, Roberts CC, Lickliter J, Krishnarajah J, Bett A, Dubey S, Finn T, Coller BA. Immunogenicity and safety of an investigational tetravalent recombinant subunit vaccine for dengue: results of a Phase I randomized clinical trial in flavivirus-naive adults. Hum Vaccin Immunother. 2019;15(9):2195-2204. doi: 10.1080/21645515.2018.1546523. Epub 2019 Jun 3. PMID 30427741
- [Result] Manoff SB, George SL, Bett AJ, Yelmene ML, Dhanasekaran G, Eggemeyer L, Sausser ML, Dubey SA, Casimiro DR, Clements DE, Martyak T, Pai V, Parks DE, Coller BA. Preclinical and clinical development of a dengue recombinant subunit vaccine. Vaccine. 2015 Dec 10;33(50):7126-34. doi: 10.1016/j.vaccine.2015.09.101. Epub 2015 Oct 14. PMID 26458804
- [Derived] Durbin AP, Pierce KK, Kirkpatrick BD, Grier P, Sabundayo BP, He H, Sausser M, Russell AF, Martin J, Hyatt D, Cook M, Sachs JR, Lee AW, Wang L, Coller BA, Whitehead SS. Immunogenicity and Safety of a Tetravalent Recombinant Subunit Dengue Vaccine in Adults Previously Vaccinated with a Live Attenuated Tetravalent Dengue Vaccine: Results of a Phase-I Randomized Clinical Trial. Am J Trop Med Hyg. 2020 Aug;103(2):855-863. doi: 10.4269/ajtmh.20-0042. Epub 2020 May 7. PMID 32394880